CLINICAL TRIAL: NCT04179318
Title: A Retrospective, International Multicenter, Single Arm Clinical Trial of the New Geneswell BCT in Vitro Diagnosis of Breast Cancer Prognosis
Brief Title: the New Geneswell BCT in Vitro Diagnosis of Breast Cancer Prognosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: The Affiliated Hospital of Hangzhou Normal University (Other); Korea University (Other)
Responsible Party: Sponsor
Other Study IDs: YANWQ002
Record Dates: First submitted 2019-10-15; First posted 2019-11-27 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- low risk: BCT Score <4
  Interventions: Diagnostic Test: Geneswell BCT
- high risk: BCT Score ≥4
  Interventions: Diagnostic Test: Geneswell BCT

INTERVENTIONS:
Diagnostic Test: Geneswell BCT — Geneswell BCT is a precise and qualitative in vitro diagnostic test. The expression of 9 genes was obtained from the formalin fixed paraffin embedded block (FFPE) of breast cancer tissue samples by RT-qPCR, and the patients were divided into high-risk group and low-risk group.

SUMMARY:
Geneswell BCT is a precise and qualitative in vitro diagnostic test. The expression of 9 genes was obtained from the formalin fixed paraffin embedded block (FFPE) of breast cancer tissue samples by RT-qPCR, and the patients were divided into high-risk group and low-risk group.

This test provides prognostic information to assess the risk of recurrence. The BCT score calculated by geneswell BCT was associated with the risk of recurrence. The higher the BCT score, the more likely it is to relapse, and vice versa.

ELIGIBILITY:
Inclusion Criteria:

* The patients were diagnosed with invasive breast cancer with positive hormone receptor (including positive estrogen receptor or progesterone receptor) and negative human epidermal growth factor receptor 2 (HER2)
* Axillary lymph node assessment : pN0 or PN1
* Women aged 18 and over
* Patients without chemotherapy after operation

Exclusion Criteria:

* Patients with negative hormone receptor （both estrogen and progesterone receptor are negative）
* Human epidermal growth factor receptor 2 （HER2） positive
* Pathological nodule evaluation: pN2 or pN3
* Male patients
* Patients receiving chemotherapy after surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with hormone receptor positive (estrogen, ER + or progesterone PR +, HER2 negative, and pN0 or PN1) early breast cancer
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2020-10-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparative assessment between risk groups | Month 9
  By evaluating the 5-year disease-free survival rate (DFS) of patients in high and low risk groups, the statistical differences between the two groups were compared.